CLINICAL TRIAL: NCT03394235
Title: Optimizing Parameters for Long-pulsed Nd:YAG Laser for Reducing Hair Shaft Diameter at the Donor Area for Hair Transplantation
Brief Title: Optimizing Parameters for Long-pulsed Nd:YAG Laser for Reducing Hair Shaft Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Dermatology, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007/2561
Record Dates: First submitted 2018-01-02; First posted 2018-01-09 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Androgenetic Alopecia; Hair Loss/Baldness
Keywords: hair transplant; hairline; laser hair removal
MeSH Terms: conditions — Alopecia | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: This is a pilot study. We plan to enroll 15 participants who requires to do hair transplantation or normal participants who are eligible for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long-pulsed, 1064nm Nd-YAG laser (Experimental): All participants will receive long-pulsed, 1064nm Nd-YAG laser treatments with three different parameters at the occipital area.
  Interventions: Device: Long-pulsed, 1064nm Nd-YAG laser

INTERVENTIONS:
Device: Long-pulsed, 1064nm Nd-YAG laser — This long-pulsed Nd-YAG laser is commonly used for laser hair removal and vascular lesions, but in this study it is used to reduce the size of the hair shaft at the occipital area.

SUMMARY:
This study evaluates the optimizing parameters of long pulse Nd:YAG Laser for reducing the size of hair shaft diameter of the donor for hair transplantation. All participants will receive long-pulsed Nd-YAG laser treatments with three different parameters at the occipital area.

DETAILED DESCRIPTION:
Since the beginning of hair transplantation era, hair transplant technique has been greatly improved to achieve the best natural looking of hairline and hair density. Most Asians tend to have large size of hair shaft at the donor area, which often cause unnatural look of the hairline at the frontal area after hair transplantation due to the contrast between the transplanted hair and the original hair.

The idea of reducing the size of the hair shaft in the certain part of donor area before being transplanted to the frontal hairline becomes appealing. This transection is being practiced extensively in the field of cosmetic medicine by using long-pulsed Neodymium-Doped:Yttrium Aluminum Gamet (Nd:YAG), a laser treatment for permanent hair removal and vascular lesions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 25-60 years with AGA or healthy
* Completed informed consent form

Exclusion Criteria:

* Pregnancy or breastfeeding
* Acute infection on the scalp or any systemic infection
* Immunocompromised host
* Chronic wasting diseases
* Use of any medications which may affect hair loss such as anticoagulants, anti-hypertensive, hormones, anticonvulsants, retinoid, mood stabilizers and antidepressants
* Unstable medical problems which may affect hair loss such as thyroid diseases, autoimmune diseases, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, congestive heart failure, cerebrovascular accident and psychiatric problems
* Hair thinning at the occipital area

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Evaluate the changes in hair density at the treated sites. | 24 weeks
  Evaluate changes in hair density at the treated sites following long-pulsed, 1064 Nd-YAG laser sessions every 8 weeks or until the treatment endpoint is reached before or at 24 weeks.

SECONDARY OUTCOMES:
Evaluate the changes in hair diameter at the treated sites. | 24 weeks
  Evaluate the changes in hair diameter at the treated sites following long-pulsed, 1064 Nd-YAG laser sessions every 8 weeks or until the treatment endpoint is reached before or at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Chinmanat Tangjaturonrusamee, MD, Study Director — Institute of Dermatology
Locations (1):
- Institute of Dermatology, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not stated in participants' informed consent.